CLINICAL TRIAL: NCT06048120
Title: First-in-man Single-dose Escalation Study in a Randomized, Single-blind, Placebo-controlled, Group-comparison Design to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BAY 2701250 After Single Short-time Intravenous Infusion or Subcutaneous Administration in Healthy Male Participants.
Brief Title: A Study to Learn How Safe the Study Treatment BAY2701250 is, How it Affects the Body and How it Moves Into, Through and Out of the Body in Healthy Male Participants When a Single Amount is Given as an Injection Into the Vein (Intravenous Infusion) or Under the Skin (Subcutaneous Injection)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: 20799; 2023-503368-18-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Hypertension Due to Left Heart Disease

STUDY DESIGN:
Intervention Model Description: This study will be conducted in a single-center, single-blind, randomized, placebo-controlled, group-comparison, dose escalation design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- i.v. infusion cohorts (Experimental): Each participant will receive a single dose of study intervention, either BAY2701250 or placebo. Study intervention will be administered by means of short time i.v. infusion. Up to 8 dose steps are planned to be investigated for i.v. administration.
  Interventions: Drug: BAY2701250 IV; Drug: Placebo IV
- s.c. injection cohorts (Experimental): Each participant will receive a single dose of study intervention, either BAY2701250 or placebo. Study intervention will be administered by means of s.c. injection. Up to 2 dose steps are planned to be investigated for s.c. administration.
  Interventions: Drug: BAY2701250 SC; Drug: Placebo SC

INTERVENTIONS:
Drug: BAY2701250 IV — Single does, intravenous infusion
  Arms: i.v. infusion cohorts
Drug: Placebo IV — Matching placebo for BAY2701250 IV
  Arms: i.v. infusion cohorts
Drug: BAY2701250 SC — Single dose, subcutaneous injection will be administered into abdominal subcutaneous fat tissue
  Arms: s.c. injection cohorts
Drug: Placebo SC — Matching placebo for BAY2701250 SC
  Arms: s.c. injection cohorts

SUMMARY:
Researchers are looking for a better way to treat people who have pulmonary hypertension (PH) due to left heart disease. PH due to left heart disease is a condition of high blood pressure in the vessels of the lungs caused by diseases in the left side of the heart.

The study treatment, BAY2701250 is under development and will be tested in humans for the first time in this study. Once it is approved, it may help treat people with PH due to left heart disease.

The participants of this study will be healthy and will have no benefit from the administration of BAY2701250. However, the study will provide important information for the design of subsequent studies with BAY2701250 in people with PH due to left heart disease. The participants will be randomly (by chance) assigned to receive either placebo or BAY2701250 as an injection into the vein (intravenous infusion) or under the skin (subcutaneous injection). A placebo is a treatment that looks like a medicine but does not have any medicine in it.

The main purpose of this first in human study is to learn how safe is BAY2701250 and to what degree medical problems caused by it can be tolerated by the study participants after they receive a single amount (dose) either as an injection into the vein (intravenous infusion) or under the skin (subcutaneous injection)?

To answer this, the researchers will collect the number of study participants with medical problems (also called adverse events) after receiving BAY2701250 until the end of the study. Doctors keep track of all adverse events that happen in studies, even if they do not think they might be related to the study treatment.

Further objectives of this study are to learn how does a single dose of BAY2701250 move into, through and out the body of the participants after an intravenous infusion or a subcutaneous injection?

To answer this, the researchers will measure:

* The (average) total level of BAY2701250 in the blood (also called AUC)
* AUC divided by dose (also called AUC/D)
* The (average) highest level of BAY2701250 in the blood (also called Cmax)
* Cmax divided by dose (Cmax/D) after receiving either an intravenous infusion or subcutaneous injection of BAY2701250.

A group of participants will start out by receiving a low dose of BAY2701250. The study doctors will look at the results from these participants and then decide whether to increase the dose of BAY2701250 in the next group of participants.

Each participant will be in the study for approximately 9-10 weeks, including a first test (screening) phase, an in-house stay of a maximum of 14 days and a follow-up phase after the end of treatment.

One visit to the study site is planned during the screening phase, followed by 6 visits (two of which are optional) after the end of treatment.

During the study, the study team will, among other:

* take blood and urine samples
* do physical examinations
* examine heart health using electrocardiogram (ECG) and
* check vital signs such as blood pressure, heart rate and body temperature

ELIGIBILITY:
Inclusion Criteria:

* Male, white participants aged 18 to 45 years
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, ECG and vital signs
* Body weight ≥ 70 kg and ≤ 100 kg as well as body mass index (BMI) within the range of 18.0 to 29.9 kg/m^2 (inclusive)
* The informed consent must be signed before any study specific tests or procedures are done
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* Medical disorder, condition, or history of such that would impair the participant's ability to participate or complete this study in the opinion of the investigator
* Thyroid disorders as evidenced by assessment of thyroid-stimulating hormone levels outside the normal reference range and confirmed by triiodothyronine and thyroxine at screening
* Known hypersensitivity to the study interventions (active substances or excipients of the preparations)
* Relevant diseases within the last 4 weeks prior to the administration of study intervention
* Febrile illness within 1 week before the administration of study intervention
* Tendency for vasovagal reactions (e.g., after venipuncture) or history of syncope
* Regular use of medicines
* Use of any drug within 14 days before the administration of study intervention, except single doses of paracetamol, ibuprofen or topical medicines
* Previous (within 90 days before first administration of study intervention) or concomitant participation in another clinical study with study intervention(s)
* Clinically relevant findings in the physical examination
* Clinically relevant findings in the electrocardiogram (ECG)
* Systolic BP below 100 or above 140 mmHg at screening for all cohorts except for the additional optional Dose Step 8 (Cohort 8) for which systolic BP below 110 or above 140 mmHg at screening will be applicable
* Diastolic blood pressure (BP) below 60 or above 90 mmHg at screening
* Pulse rate below 50 or above 90 beats per minute at screening
* Positive urine drug screening
* Positive alcohol breath test
* Positive results for human immunodeficiency virus (HIV) antibodies (anti-HIV 1+2), or HIVp24 antigen
* Positive results for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (anti-HCV)
* Clinically relevant deviations of the screened safety laboratory parameters in clinical chemistry, hematology, or urinalysis from reference ranges at screening
* Smoking
* Regular daily consumption of more than 1 L of methylxanthine-containing beverages
* Regular daily consumption of more than 500 mL of usual beer or the equivalent quantity of approximately 20 g of alcohol in another form
* Unable/unwilling to comply with study restrictions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | From administration of study intervention until last follow-up visit, up to 46 (+3) days after administration

SECONDARY OUTCOMES:
AUC of BAY2701250 in plasma | From pre-dose up to 77 days after i.v. administration, respectively up to 81 days after s.c. administration
  AUC: Area under the concentration vs. time curve from zero to infinity after single dose
  AUC(0-t), may be evaluated as main parameter if AUC cannot be reliably determined in all participants
AUC/D of BAY2701250 in plasma | From pre-dose up to 77 days after i.v. administration, respectively up to 81 days after s.c. administration
  AUC(0-t)/D, may be evaluated as main parameter if AUC/D cannot be reliably determined in all participants
Cmax of BAY2701250 in plasma | From pre-dose up to 77 days after i.v. administration, respectively up to 81 days after s.c. administration
  Cmax: Maximum observed drug concentration
Cmax/D of BAY2701250 in plasma | From pre-dose up to 77 days after i.v. administration, respectively up to 81 days after s.c. administration
F as ratio of the respective s.c. to i.v. values determined for AUC | From pre-dose up to 81 days after administration
  F: Absolute bioavailability

CONTACTS AND LOCATIONS:
Locations (1):
- NUVISAN GmbH Neu-Ulm, Neu-Ulm, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/20799